CLINICAL TRIAL: NCT05362786
Title: Bone Marrow-Derived Mesenchymal Stem Cell Therapy for Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LaTonya J. Hickson (Other)
Responsible Party: Sponsor-Investigator, LaTonya J. Hickson, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21-011822
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Arm 1 (Experimental): Subjects with chronic kidney disease will receive allogeneic bone marrow-derived mesenchymal stem cells (MSC) in two intravenous infusions of 100x10^6 cells at time zero and three months
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)
- Dose Arm 2 (Experimental): Subjects with chronic kidney disease will receive allogeneic bone marrow-derived mesenchymal stem cells (MSC) single intravenous infusion of 200x10^6 cells
  Interventions: Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC)

INTERVENTIONS:
Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC) — Two intravenous infusions delivered systemically through a peripheral IV(over 30 minutes to 2 hours) of 100x10^6 cells at day 0 and day 84
  Arms: Dose Arm 1
Drug: Allogeneic adipose-derived mesenchymal stem cells (MSC) — Single intravenous infusion delivered systemically through a peripheral IV(over 30 minutes to 2 hours) of 200x10^6 cells at day 0
  Arms: Dose Arm 2

SUMMARY:
The purpose of this study is to assess the safety and tolerability of intravenously delivered mesenchymal steml cells (MSC) in one of two fixed dosing regimens at two time points in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-80 years
2. Estimated glomerular filtration rate (eGFR) 25-55 ml/min/1.73m2

   1. If eGFR 45-55 ml/min/1.73m2, then albumin:creatinine ratio ≥300 mg/g or proteinuria ≥300 mg/day despite maximally tolerated dose of RAAS drugs (e.g. ACE Inhibitors, Angiotensin Receptor Blockers)
   2. If eGFR 25-44 ml/min/1.73m2, must have urine albumin:creatinine ratio ≥30mg/g despite maximally tolerated dose of RAAS drugs (e.g. ACE Inhibitors, Angiotensin Receptor Blockers)
3. Hemoglobin A1c of ≤ 8% despite maximally tolerated anti-diabetes therapy
4. Ability to give informed consent

Exclusion Criteria:

1. Anemia (hemoglobin <9 g/dL)
2. Body weight >150 kg or BMI >50
3. Uncontrolled hypertension: sustained systolic blood pressure (SBP) >150 mmHg or diastolic blood pressure (DBP) ≥100 mmHg despite maximal doses of at least 2 different classes of anti-hypertensive medications
4. Chronic hypotension history: sustained SBP <85 mmHg
5. Glomerulonephritis not in partial or complete remission for 6 months (or estimated/ measured proteinuria greater than 10 grams/day),
6. Active glomerulonephritis (glomerular diseases with evidence of active urinary sediment, serology or biopsy findings) including ANCA-associated glomerulonephritis, post-infectious glomerulonephritis, lupus nephritis, amyloidosis, or other monoclonal gammopathy of renal significance
7. Autosomal dominant or recessive polycystic kidney disease
8. Nephrotic syndrome defined as proteinuria >3.5 g per 24 hours, plus hypoalbuminemia (serum albumin less than or equal to 2.5 g/L) and edema.
9. Proteinuria >5 g/day (with or without nephrotic syndrome).
10. Kidney failure requiring renal replacement therapy (hemodialysis, peritoneal dialysis, or kidney transplantation)
11. Active immunosuppression therapy (including prednisone greater than or equal to 10 mg daily)
12. Kidney transplantation history
13. Solid organ transplantation history
14. Recent cardiovascular event (myocardial infarction, stroke, congestive heart failure (NYHA class ≥III or ejection fraction ≤30%) within 6 months or uncontrolled cardiac arrhythmias (e.g. ventricular arrhythmia, supraventricular tachycardia and bradyarrhythmia)
15. History of liver cirrhosis
16. Chronic obstructive pulmonary disease or asthma requiring daily medication
17. History of blood clotting disorder (thromboembolism; pulmonary embolism, deep venous thrombosis)
18. Pregnancy
19. Unwilling to use contraception for at least 2 months after MSC infusion if sexually active and able to become pregnant or father a child.
20. Active malignancy
21. Active infection (e.g. systemic or specific organ involvement such as pneumonia or osteomyelitis)
22. Recent COVID-19 infection within the last 3 months
23. History of hepatitis B or C (without cure), or HIV infection
24. History of allergic reaction to cellular products (ie. blood transfusions, platelets)
25. Active tobacco use
26. Illicit drug use and excessive alcohol use
27. Presence of psychosocial issues (e.g., uncontrolled mental illness, unpredictable childcare or eldercare responsibilities, irregular/ inflexible work schedule) that may interfere with the ability to complete all study procedures
28. Subjects anticipating prolonged travel or other physical restrictions that would prohibit return for scheduled study visits.
29. Inability to give informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Adverse events and/or serious adverse events | 15 months
  Number of adverse events and/or serious adverse events associated with mesenchymal stem cells intervention
Change in eGFR Value | 6 months
  Blood serum estimated glomerular filtration rate (eGFR) reported in milliliters per minute (mL/min)

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya Hickson, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Patel HA, Wang J, Zinn CJ, Learmonth M, Lerman LO, Wolfram J, Hickson LJ. Fortifying the Diabetic Kidney Disease Treatment Armamentarium: Multitarget Senotherapeutic and Regenerative Strategies. J Am Soc Nephrol. 2025 May 7;36(8):1655-1658. doi: 10.1681/ASN.0000000754. No abstract available. PMID 40333016
- [Derived] Andrews TD, Day GS, Irani SR, Kanekiyo T, Hickson LJ. Uremic Toxins, CKD, and Cognitive Dysfunction. J Am Soc Nephrol. 2025 Jun 1;36(6):1208-1226. doi: 10.1681/ASN.0000000675. Epub 2025 Feb 26. PMID 40009460
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials